CLINICAL TRIAL: NCT04784182
Title: Synbiotic Supplementation to Reduce Anxiety Symptoms in Female Breast Cancer Survivors and/or Their Female Relatives
Brief Title: Anti-anxiety Biotics for Breast Cancer Survivors
Acronym: ABBCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only three participants enrolled
Sponsor: Auburn University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Andrew Fruge, Assistant Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 21-110; UL1TR003096-03 (NIH)
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Anxiety Generalized; Breast Cancer Female
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Placebo controlled randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: One study staff member will be responsible for randomization and allocation of intervention supplement or placebo, which will be appear to be identical
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic supplement group (Experimental): Daily consumption of pills containing prebiotics and probiotics
  Interventions: Dietary Supplement: probiotic plus prebiotic supplement
- Placebo group (Placebo Comparator): Daily consumption of pills containing maltodextrin
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotic plus prebiotic supplement — Daily consumption of probiotic containing at least 5 billion CFU per day total bacteria including Lactobacillus helveticus and Bifidobacterium longum and prebiotic containing 4 grams of fructooligosaccharides (FOS)
  Arms: Synbiotic supplement group
Dietary Supplement: placebo — Daily consumption of visually similar placebo pills
  Arms: Placebo group

SUMMARY:
Cancer survivors experience more rapid declines in health-related quality of life which include physical and psychological comorbidities, the latter of which may be subclinical and often overlooked by primary care providers. Recently, the gut-brain axis (GBA) has been identified as a therapeutic target to improve host health. The GBA is greatly influenced by the composition of the gut microbiome, as microbial metabolites directly influence the central nervous system. Thus, prebiotics, probiotics, and synbiotics (a combination of pre- and probiotics) have emerged as a possible approach to treating anxiety symptoms. Preclinical studies suggest efficacy of synbiotics, while pre- and probiotics have only been studied in isolation in humans.

This is a double-blind, placebo-controlled clinical trial in which female breast cancer survivors and/or their female relatives experiencing moderate to severe anxiety symptoms will be randomized to daily consumption of the synbiotic supplement or placebo. The previously validated Generalized Anxiety Disorder-7 (GAD-7) will be used to assess anxiety symptom severity at study screening and at each time point. The primary outcome of this study is feasibility, measured by accrual, adherence, retention, and adverse effects. Secondary outcomes relate to reduction of anxiety symptoms and other physiological changes. No study has investigated the mediating effects of gut microbiota and inflammatory markers on the ability of synbiotics to reduce anxiety symptoms. Thus, at each timepoint, phlebotomy will be conducted to determine serum levels of inflammatory cytokines and stool samples will be collected to determine alpha- and beta-diversity of the fecal microbiome as well as relative abundance of target genera. Hypothesis: this placebo-controlled study will be feasible and synbiotic treatment will result in a significant reduction in anxiety symptoms and inflammatory markers, which may be moderated by changes in the microbiome.

ELIGIBILITY:
Inclusion Criteria:

Female breast cancer survivors or female relatives of a breast cancer survivor who:

1. are 50 years of age or older
2. have completed primary treatment
3. currently experience clinical anxiety symptoms determined by the 7 item Generalized Anxiety Disorder screener (GAD-7; eligibility requires a total score of 5 or higher on the 21 point scale)
4. agree not to change dietary supplements throughout the course of the study
5. are willing to comply with daily supplement regimen
6. are able to speak and read English.

Exclusion Criteria:

1. use of any of the following drugs within the last 4 weeks (unless indefinitely prescribed): systemic antibiotics, corticosteroids, immunosuppressive agents, or commercial probiotics
2. changes in treatment for anxiety symptoms (i.e. initiation of Cognitive Behavior Therapy (CBT) within the last four weeks
3. current use (within 12 weeks) of anxiolytic medications.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Frugé, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith KS, Greene MW, Babu JR, Fruge AD. Psychobiotics as treatment for anxiety, depression, and related symptoms: a systematic review. Nutr Neurosci. 2021 Dec;24(12):963-977. doi: 10.1080/1028415X.2019.1701220. Epub 2019 Dec 20. PMID 31858898
- See also: Study website — http://aub.ie/survivor

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No pre-assignment activities. Participants were randomized and received intervention or treatment immediately after baseline data collection was completed.
Period: Overall Study
Arm/Group | Synbiotic Supplement Group | Placebo Group
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synbiotic Supplement Group | Placebo Group | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 55 [55 to 55] | 62.5 [58 to 67] | 60 [55 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3
Generalized Anxiety Disorder Screener (GAD-7) Score [Mean (Standard Deviation); unit: units on a scale (min=0; max=21)] — 7 items, 0-3 score for each response; 21 points possible - Range 0-21. No subscales. Higher score is a less desirable outcome.
  units on a scale (min=0; max=21) | 8 | 8 (4.24) | 8 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Accrual
Description: Number of Participants who were accrued in 6 months
Time Frame: 6 months
Population: Number of Participants who were accrued in 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Synbiotic Supplement Group | Placebo Group
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

2. Primary Outcome: Feasibility - Retention
Description: Retain 85% of randomized participants for duration of study (6 weeks)
Time Frame: 6 weeks
Population: All participants analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Synbiotic Supplement Group | Placebo Group
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

3. Primary Outcome: Feasibility - Adherence
Description: 80% of participants consuming pills on 90% of intervention days
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Synbiotic Supplement Group | Placebo Group
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

4. Secondary Outcome: Anxiety Symptoms
Description: Decrease in Generalized Anxiety Disorder-7 (GAD-7) score, which ranges from 0 (no anxiety) to 21 (severe anxiety).
Time Frame: 4 weeks
Population: Outcome cannot be reported. Identification of age and race in baseline characteristics with total sample of n=3 compromises personally identifiable information.
Arm/Group | Synbiotic Supplement Group | Placebo Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Serotonin
Description: Serum 5-hydroxytryptamine
Time Frame: 4 weeks
Population: Biospecimen samples will never be analyzed. Data not collected.
Arm/Group | Synbiotic Supplement Group | Placebo Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Inflammatory Marker - TNF-alpha
Description: Serum Tumor Necrosis Factor-alpha
Time Frame: 4 weeks
Population: Biospecimen samples will never be analyzed. Data not collected.
Arm/Group | Synbiotic Supplement Group | Placebo Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Inflammatory Marker - LBP
Description: Serum Lipopolysaccharide Binding Protein
Time Frame: 4 weeks
Population: Biospecimen samples will never be analyzed. Data not collected.
Arm/Group | Synbiotic Supplement Group | Placebo Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Inflammatory Marker - IL-6
Description: Pro-inflammatory cytokine, Interleukin-6 (serum)
Time Frame: 4 weeks
Population: Biospecimen samples will never be analyzed. Data not collected.
Arm/Group | Synbiotic Supplement Group | Placebo Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Fecal Microbiome Composition
Description: 16s changes in microbiota alpha diversity
Time Frame: 4 weeks
Population: Biospecimen samples will never be analyzed. Data not collected.
Arm/Group | Synbiotic Supplement Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Synbiotic Supplement Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
Biospecimen samples will never be analyzed. Data not collected for secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT04784182/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT04784182/ICF_001.pdf